CLINICAL TRIAL: NCT04746378
Title: Comparison of Predictive Value of Different Stone Burden Measurements for Outcomes After Urinary Stone Treatment.
Brief Title: PRedictive Accuracy of Initial Stone Burden Evaluation.
Acronym: PRAISE
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: EAU Young Academic Urologists Urolithiasis and Endourology Working Group (Unknown); European Association of Urology Section of Uro-Technology (Unknown); Endourological Society TOWER Research Team (Unknown)
Responsible Party: Sponsor
Other Study IDs: BC-7295
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Urolithiasis; Ureterolithiasis; Nephrolithiasis
Keywords: ureteroscopy; extracorporeal shockwave lithotripsy; percutaneous nephrolithotomy; stone burden; non-contrast computed tomography
MeSH Terms: conditions — Urolithiasis; Ureterolithiasis; Nephrolithiasis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- extracorporeal shockwave lithotripsy: Patients that are included in the study and undergo a shockwave lithotripsy. The pre- and postoperative assessment remains the same across groups
  Interventions: Diagnostic Test: Computed Tomography, CSD; Diagnostic Test: Computed Tomography, SA; Diagnostic Test: Computed Tomography, 3D
- uretero(reno)scopy: Patients that are included in the study and undergo a semirigid or flexible uretero(reno)scopy. The pre- and postoperative assessment remains the same across groups
  Interventions: Diagnostic Test: Computed Tomography, CSD; Diagnostic Test: Computed Tomography, SA; Diagnostic Test: Computed Tomography, 3D
- percutaneous nephrolithotomy: Patients that are included in the study and undergo a percutaneous nephrolithotomy. The pre- and postoperative assessment remains the same across groups
  Interventions: Diagnostic Test: Computed Tomography, CSD; Diagnostic Test: Computed Tomography, SA; Diagnostic Test: Computed Tomography, 3D

INTERVENTIONS:
Diagnostic Test: Computed Tomography, CSD — Measurement of the stone burden by cumulative stone diameter, the sum of linear longest diameters of all the stones to be treated within one patient as measured on the CT or by additional rendering software
  Other Names: Cumulative Stone Diameter
Diagnostic Test: Computed Tomography, SA — Measurement of the stone burden by surface area, the sum of surface areas of all the stones to be treated within one patient as measured on the CT or by additional rendering software
  Other Names: Stone Surface Area
Diagnostic Test: Computed Tomography, 3D — Measurement of the stone burden by volume of all the stones to be treated within one patient, as measured on the CT or by additional rendering software
  Other Names: Stone Volume

SUMMARY:
This study is intended to be a prospective registry of patients undergoing any kind of stone treatment that have a pre-operative CT available. This imaging will be used to measure the stone burden in three different ways: in a single dimension (cumulative stone diameter), in two dimensions (surface area) and in three dimensions (volume).The primary purpose is to identify what way of measuring stone burden is most predictive of outcomes after stone treatment such as stone free status, operative time and complications.

DETAILED DESCRIPTION:
The current EAU and AUA guidelines still base the recommendations for stone treatment on cumulative stone diameter, a linear measurement of the stone burden. Multiple nomograms rather use the stone burden's surface area to predict post-operative outcomes. More recently, volume has been prposed as the most accurate measure of stone burden and the variable to be reported in stone treatment literature. Although inuitively a three dimensional evaluation is most likely the most accurate representation of the stone burden to be treated.

Several reports however have compared different ways of measuring stone burden and could not confidently identify volume as the most accurate predictor of surgical outcomes.

With this study, we aim to prospectively collect data on a large group of patients that have a pre-operative CT scan available. This imaging will be used to assess the stone burden in different ways, linear, two dimensional and three dimensional. Both procedural and post-operative data will be collected to identify which of the measurements is most accurate in predicting outcomes such as stone free status, operative time and complications such as bleeding. Patients can be included regardless of the procedure that is proposed to treat the stone. After inclusion and after having undergone the procedure, at least one post-operative assessment is necessary to be able to evaluate the pre-operative variables against post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Availability of computed tomography imaging
* Undergoing any of the previously described procedures: extracorporeal shockwave lithotripsy, uretero(reno)scopy or percutaneous nephrolithotomy
* Able to read and understand the information regarding the study and able to provide informed consent

Exclusion Criteria:

* Under the stated age limit
* No pre-operative computed tomography imaging available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing any stone treatment that have a pre-operative CT that can be used for post-processing evaluation of the stone burden with specified software. Primary stone treatment only.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Stone Free Status | 1 day to 3 months
  Any residual stone fragments after the initial treatment

SECONDARY OUTCOMES:
Operative Time | intra-operative
  Time needed to treat the stone burden as measured during one treatment session
Complication | 30 days
  Any complication thet can be attributed to the procedure that was performed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tailly, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Eastern-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Currently, we have not planned to share individual patient data with any other researchers